CLINICAL TRIAL: NCT05672823
Title: Minimally-Invasive Upper Extremity Approach Versus Lower Extremity Approach for Transcatheter Aortic Valve Implantation (TAVI) Accessory Access Sites; A Prospective, Multicenter, Investigator-Initiated, Randomized Clinical Trial
Brief Title: Upper Extremity Versus Lower Extremity Accessory Access Sites During Transcatheter Aortic Valve Implantation
Acronym: TAVIXS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL80895.091.22
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Coronary angiography; Hemorrhage; Hospitalization; Pacemaker
MeSH Terms: conditions — Aortic Valve Stenosis; Hemorrhage | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor, being the trial statistician, is blinded for the treatment groups.
  Groups are defined as group A and B during the preparation of the statistical tests. Only after performing the required statistical tests the data will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive, upper extremity (Experimental): Radial artery for pigtail catheter and pacing over the Left Ventricular (LV) stiff wire OR radial artery for pigtail catheter and brachial vein for temporary pacemaker when not pacing over the LV stiff wire.
  Interventions: Procedure: Transcatheter Aortic Valve Implantation (TAVI)
- Lower extremity (Active Comparator): Femoral artery for pigtail catheter and pacing over the LV stiff wire OR femoral artery for pigtail catheter and femoral vein for temporary pacemaker when not pacing over the LV stiff wire.
  Interventions: Procedure: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation (TAVI) — Comparing different accessory access sites for TAVI: the temporary pacemaker access site and the diagnostic access site.

SUMMARY:
The goal of this prospective, multicenter, investigator-initiated, randomized clinical trial is to assess the safety and efficacy of a 'minimally invasive, upper extremity' approach versus the standard 'lower extremity' approach for accessory access sites in patients undergoing a transcatheter aortic valve implantation.

The main questions it aims to answer are whether a 'minimally invasive, upper extremity' approach as compared with the standard 'lower extremity' approach:

* Is associated with less clinically relevant access site-related bleeding complications.
* Is associated with a shorter time to mobilization after TAVI.
* Is associated with a shorter duration of hospitalization.
* Has the same early safety outcomes at 30 days post-TAVI.

Participants will be subject to the usual care surrounding a TAVI procedure but will also will be asked to fill out two questionnaires before and after TAVI:

* Quick Disabilities of the Arm, Shoulder and Hand (Quick DASH)
* Lower Extremity Functional Scale (LEFS)

Researchers will compare the minimally invasive, upper extremity group with the standard lower extremity to see if there are difference regarding the posed questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 18 years old.
* Written informed consent is obtained from all patients.
* Planned for transfemoral TAVI procedure.

Exclusion Criteria:

* Inability to obtain informed consent.
* Contra-indication for brachial or femoral vein access (temporary pacemaker access site).
* Contra-indication for radial or femoral artery access (diagnostic access site).
* Use of a cerebral embolic protection device (CEPD) if this requires an additional (arterial) access site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Clinically relevant bleeding of the randomized access site; either diagnostic or pacemaker access site, or both | "Through 30 days"
  Bleeding Academic Research Consortium (BARC) type 2, 3 or 5 bleeding; In case a clinically relevant bleeding occurs in both the randomized diagnostic access site and the randomized pacemaker access site, these will be combined and the highest classification of the two BARC bleedings will be scored.
  BARC classification: a classification scoring bleeding complication based on the clinical actions that follow in which type 1 bleeding is not actionable and type 5 bleeding is fatal.

SECONDARY OUTCOMES:
Time to mobilization | "during index hospitalization, approximately 3 days - often hours after TAVI procedure"
  Time to first mobilization in minutes after procedure; mobilization is defined as walking short distances on the patients room or on the corridor. Transfers between bed and chair are not measured as mobilization.
Total duration of hospitalization | "during index hospitalization, approximately 3 days"
  Duration of index hospitalization in days.
Composite endpoint of all clinically relevant bleeding of the access sites; either diagnostic or pacemaker access site or primary (TAVI) access site | "Through 30 days"
  Bleeding Academic Research Consortium (BARC) type 2, 3 or 5 bleeding of either the diagnostic access, pacemaker access or primary (TAVI) access.
Clinically relevant bleeding not related to the randomized access sites | "Through 30 days"
  Bleeding Academic Research Consortium (BARC) type 2, 3 or 5 bleeding not related to the diagnostic access or pacemaker access.
All-cause mortality | "30 days"
  Deaths within the first 30 days after procedure from any cause.
All stroke | "30 days"
  All cerebrovascular accidents within the first 30 days after procedure.
Valve Academic Research Consortium-3 (VARC) type 2-4 bleeding | "30 days"
  Bleeding criteria following the VARC-3 criteria. Type 2 bleeding is classified as bleeding requiring transfusion. Type 3 bleeding is defined as bleeding in a critical organ, causing hypovolemic shock, requiring reoperation or significant transfusion.
  Type 4 bleeding is defined as overt bleeding leading to death.
Major vascular, access-related, or cardiac structural complications | "30 days"
  Major vascular complications:
  * Aortic dissection or aortic rupture.
  * Vascular (arterial or venous) injury, unplanned endovascular or surgical intervention, closure device failure, distal embolization or compartment syndrome resulting in death, VARC type ≥ 2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment.
  Major access-related complications:
  • Non-vascular structure, non-cardiac structure perforation, injury, or infection resulting in death, VARC type ≥ 2 bleeding, irreversible nerve injury or requiring unplanned surgery or percutaneous intervention
  Major cardiac structural complications:
  • Cardiac structure perforation, injury, new pericardial effusion, coronary obstruction or compromise resulting in death,VARC type ≥ 2 bleeding, haemodynamic compromise or tamponade, or requiring unplanned surgical or percutaneous intervention.
Acute kidney injury stage 3 or 4 | "30 days"
  All cases of acute kidney injury stage 3 or 4 within 30 days after procedure.
Moderate or severe aortic regurgitation | "30 days"
  All cases of moderate or severe aortic regurgitation within 30 days after procedure.
New permanent pacemaker due to procedure-related conduction abnormalities | "30 days"
  All permanent pacemaker placements in the first 30 days after procedure due to procedure-related conduction abnormalities.
Surgery or intervention related to the device | "30 days"
  All cases of surgery or interventions related to the device within 30 days after procedure.

OTHER OUTCOMES:
Frequency rate of cross-over to the non-randomized access site | "Immediately after procedure"
  Frequency rate of cross-over of either the diagnostic or temporary pacemaker access site, or both.
Fluoroscopy time | "Immediately after procedure"
  Fluoroscopy time during the procedure measured in minutes.
Skin-to-skin time | "Immediately after procedure"
  Skin-to-skin time of the total procedure measured in minutes.
Number of punctions for diagnostic access | "Immediately after procedure"
  The number of punctions before secondary arterial (diagnostic) access was achieved.
Number of punctions for temporary pacemaker access | "Immediately after procedure"
  The number of punctions before temporary pacemaker access was achieved.
Temporary pacemaker failure | "during index hospitalization, approximately 3 days"
  Defined as either:
  * Failure to capture
  * Failure to pace
  * Failure to sense intrinsic beats
Pacemaker lead in situ duration | "during index hospitalization, approximately 3 days"
  The duration for which the temporary pacemaker wire was in situ in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Niels van Royen, prof. dr., Principal Investigator — Radboud University Medical Center
Locations (8):
- Netherlands (8):
  - Radboud university medical center, Nijmegen, Gelderland
  - Amsterdam UMC, Amsterdam
  - OLVG, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht UMC, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Isala Zwolle, Zwolle

REFERENCES:
- [Derived] Versteeg GAA, Rooijakkers MJP, Hemelrijk KI, Vlaar PJ, Overduin DC, van Wely MH, Aarts HM, van Ginkel DJ, Stens NA, van Nunen LX, van Geuns RJ, van Garsse LAFM, Geuzebroek GSC, Verkroost MWA, Cetinyurek-Yavuz A, Heijmen RH, Thijssen DHJ, Ten Berg JM, Tonino PAL, Delewi R, van Royen N. Extremity Function After Transfemoral Transcatheter Aortic Valve Implantation: A TAVI XS Sub-Study. Catheter Cardiovasc Interv. 2026 Jan 13. doi: 10.1002/ccd.70470. Online ahead of print. PMID 41527810
- [Derived] Versteeg GAA, Rooijakkers MJP, Hemelrijk KI, Vlaar PJ, Overduin DC, van Wely MH, Aarts HM, van Ginkel DJ, van Nunen LX, van Geuns RJ, van Garsse LAFM, Geuzebroek GSC, Verkroost MWA, Cetinyurek-Yavuz A, Heijmen RH, Ten Berg JM, Tonino PAL, Delewi R, van Royen N. Upper- vs Lower-Extremity Secondary Access During Transcatheter Aortic Valve Implantation: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2438578. doi: 10.1001/jamanetworkopen.2024.38578. PMID 39412806